CLINICAL TRIAL: NCT05607901
Title: A Comparative Clinical Trial Evaluating the Effect and Safety of Tacrolimus Versus Hydrocortisone in Management of Atopic Dermatitis in Children
Brief Title: A Comparative Clinical Trial Evaluating the Effect and Safety of Tacrolimus Versus Hydrocortisone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35928
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Dermatologic Disease
MeSH Terms: conditions — Skin Diseases | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: • A randomized, controlled, and parallel study will comprise 100 patients with AD
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus Group (Active Comparator): 50 patients will be treated with a thin layer of 0.03% topical tacrolimus ointment on the affected areas twice daily for 4 months.
  Interventions: Drug: Tacrolimus ointment
- Hydrocortisone Group (Active Comparator): 50 patients will be treated with a thin layer of 1% hydrocortisone cream on the affected areas twice daily for 4 months.
  Interventions: Drug: Hydrocortisone 1% cream

INTERVENTIONS:
Drug: Tacrolimus ointment — tacrolimus is an immunosuppressive drug acting as an immunomodulator to assist manage acute flares and reducing the severity of future flares
  Arms: Tacrolimus Group
Drug: Hydrocortisone 1% cream — Topical corticosteroids (TCS) are the cornerstone for the management of AD to which other treatments are compared.
  Arms: Hydrocortisone Group

SUMMARY:
One of the most frequent skin conditions is atopic dermatitis (AD), characterized by its pruritic inflammation effect. Where the prevalence of AD increased in the last three decades by two or three folds worldwide, especially in developed countries, AD is supposed to affect about 15% to 30% of children, and 2% to 10% of adults. This type of dermatitis is frequently linked to a family history of other atopic illnesses such as allergic rhinitis or asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 2-16 years old AD patients.

Exclusion Criteria:

* patients diagnosed with other skin disorders of serious type and who are taking systemic corticosteroids or anti-inflammatory medications.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
To compare the impact of topical tacrolimus ointment to topical hydrocortisone cream by measuring inflammatory cytokine levels in the blood. | 4 months
  To compare the impact of topical tacrolimus ointment to topical hydrocortisone cream by measuring inflammatory cytokine levels in the blood such as interleukin-6 (IL-6), and IL-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt

REFERENCES:
- [Derived] Binsaleh AY, Bahaa MM, Elmasry TA, Elberri EI, Kotkata FA, El-Khateeb E, Kamal M, El-Samongy MA, Hamouda AO, Alghamdi AM, Alrubia S, Salahuddin MM, Eltantawy N. A randomized controlled trial comparing tacrolimus versus hydrocortisone for the treatment of atopic dermatitis in children: new perspectives on interferon gamma-induced protein and growth-related oncogene-alpha. Front Med (Lausanne). 2024 Jul 24;11:1399305. doi: 10.3389/fmed.2024.1399305. eCollection 2024. PMID 39114823